CLINICAL TRIAL: NCT01400672
Title: Imiquimod/BTIC Lysate-Based Vaccine Immunotherapy for Diffuse Intrinsic Pontine Glioma in Children and Young Adults
Brief Title: Imiquimod/Brain Tumor Initiating Cell (BTIC) Vaccine in Brain Stem Glioma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Treatment ineffective; Extreme toxicity
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009LS136; 1004M81213 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2011-07-19; First posted 2011-07-22 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Diffuse Intrinsic Pontine Glioma
Keywords: Diffuse intrinsic pontine glioma
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma | interventions — Imiquimod; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DIPG Patients Receiving Vaccine (Experimental): Patients with diffuse intrinsic pontine glioma (DIPG) receiving radiation therapy, Tumor Lysate Vaccine (dose of 4 x 10^6 cells divided into 2 doses then every 4 weeks for up to 1 year) and Imiquimod (5% Aldara cream at a total dose of 12.5 mg) topically at each site prior to and 24 hours after vaccination.
  Interventions: Biological: Tumor Lysate Vaccine; Drug: Imiquimod; Radiation: Radiation therapy

INTERVENTIONS:
Biological: Tumor Lysate Vaccine — Vaccination is injected intradermally every 2 weeks for 4 doses, then every 4 weeks for up to 1 year. Patients will receive 1 mg protein divided into 2 doses at two separate subinguinal sites.
Drug: Imiquimod — Marketed as 5% Aldara cream topically applied; total of 12.5 mg divided between the two vaccination sites and reapplied at the vaccination sites 24 hours later.
  Other Names: Aldara cream
Radiation: Radiation therapy — Initial course of radiation therapy is given over 6-7 weeks, 5580 cGy. At the time of the 3rd vaccination, an additional 180 cGy fractions will be delivered in single doses in a novel effort to induce NKG2D ligand upregulation (thereby "sensitizing" residual tumor to lymphocyte attack). The total radiation dose for each patient will be 5760 cGy.

SUMMARY:
This is a pilot/feasibility study. The study design represents a modification of current standard of care for Diffuse Intrinsic Pontine Glioma (DIPG) (5580 cGY involved field radiation), with the final two doses of radiation given at intervals during the vaccination phase of treatment.

Patients between the ages of 3 years and 25 years diagnosed with Diffuse Intrinsic Pontine Glioma (DIPG) will be allowed to participate in the trial. Study enrollment will occur after the completion of conformal radiation therapy to a dose of 5580 cGy and the post radiation therapy (RT) magnetic resonance imaging (MRI) shows no disease progression.

Three patients with glioblastoma multiforme, aged 16 years and older, will be entered first to confirm vaccine safety before enrolling DIPG patients.

DETAILED DESCRIPTION:
Vaccine will be produced by the University Of Minnesota Molecular and Cellular Therapeutics Facility using the established brain tumor initiating cell (BTIC) cell line GBM-6 as the antigen source. Vaccine administration will begin at four weeks (week 10) following completion of radiation therapy and will be given every two weeks for four doses. At the time of the 1st and 3rd vaccinations, additional 180 cGy fractions will be delivered in single doses in a novel effort to induce NKG2D ligand upregulation (thereby "sensitizing" residual tumor to lymphocyte attack). The total radiation dose for each patient will be 5940 cGy. Subsequent vaccinations will be given every four weeks and will continue to a maximum of one year from study enrollment, by which time median survival will have passed based on historical data. Imaging will be obtained at study entry (post radiation therapy) and every eight weeks thereafter to eighteen months, after which time the interval between imaging follow-up episodes will be determined by the patient's clinical status. Imaging will include MRI of the brain using our current institutional brain tumor imaging protocol. Imaging will also include SPECT/MRI and perfusion MRI. FDG-PET imaging may be used in certain cases to differentiate tumor necrosis from progression.

ELIGIBILITY:
Inclusion Criteria

* Age 16 years or older patients with histologically confirmed glioblastoma multiforme (GBM) World Health Organization (WHO) grade III-IV with recurrent or progressive disease after standard therapy (enrollment plan 1).
* Age 3 years and older patients with diffuse intrinsic pontine glioma (DIPG) diagnosed by magnetic resonance imaging (MRI). Completion of standard radiation therapy (not to exceed 5580 cGy) with a post radiation therapy (RT) MRI that shows no disease progression when compared with pre-RT MRI. All patients must be treated with Intensity Modulated Radiation Therapy (IMRT) or an equivalent conformal technique. Patients from an outside institution who are referred after the start of radiation therapy may complete initial radiation therapy at their home institution as long as dosage guidelines are met and the total dose does not exceed 5580 cGy at the time of study registration (enrollment plan 2 and 3).
* all patients regardless of diagnosis must be clinically stable and off or on low dose (no more than 0.1 mg/kg/day, maximum of 4 mg/day dexamethasone) corticosteroid for at least 1 week prior to study enrollment.

Exclusion Criteria:

* Pregnant or breast-feeding. Pregnancy testing will be performed on all menstruating females within 14 days prior to study enrollment.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements
* Currently receiving any chemotherapy, investigational agents or registration on another therapy based trial or received chemotherapy with radiation therapy
* History of immune system abnormalities such as hyperimmunity (e.g., autoimmune diseases) and hypoimmunity (e.g., myelodysplastic disorders, marrow failures, AIDS, ongoing pregnancy, transplant immunosuppression)
* Any isolated laboratory abnormality suggestive of a serious autoimmune disease
* Any conditions that could potentially alter immune function (AIDS, multiple sclerosis, diabetes, renal failure)
* Receiving ongoing treatment with immunosuppressive drugs, excluding those patients requiring dexamethasone for treatment of tumor-related edema

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-07-17 (Actual); Primary Completion 2016-03-07 (Actual); Study Completion 2018-10-08 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity | Within 24 hours of vaccination
  Determined as Grade 3 or 4 toxicity observation after dosing with BTIC vaccination. Toxicity will be graded using the NCI's Common Terminology Criteria for Adverse Events (CTCAE 4.0) in terms of local, regional and systemic events.

SECONDARY OUTCOMES:
Time to Tumor Progression | Study entry through 24 months after treatment
  Imaging will include MRI, SPECT/MRI and perfusion MRI. FDG-PET imaging may be also be used Response criteria: Complete responses (CR) are those in which there is a disappearance of all enhancing tumor or tumor mass on consecutive MRI scans. Patients must be off steroids, and neurologically stable or improved.
  Partial responses (PR) are those in which there is a ≥ 50% reduction in the size of the enhancing tumor or tumor mass on consecutive MRI scans. In addition, the patient must be neurologically stable.
Drop-out rate | 24 hours, 48 hours and 1 week after each vaccination
  Treatment feasibility will be based on the drop-out rate in absence of disease progression. Information will be presented in a tabular and descriptive manner

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Moertel, M.D., Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States